CLINICAL TRIAL: NCT07149922
Title: Early Blood Pressure Intervention After Coiling or Clipping for Subarachnoid Hemorrhage
Acronym: EPIC-SAH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Development Center for Medical Science & Technology National Health Commission of the People's Republic of China (Unknown); Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Xiaolin Chen, MD, Early Blood Pressure Intervention after Coiling or Clipping for Aneurysmal Subarachnoid Hemorrhage, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2024-267-01; 2023ZD0505106 (Other Grant/Funding Number: Development Center for Medical Science & TechnologyNational Health Commission of the People's Republic of China)
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Aneurysmal Subarachnoid Hemorrhage (aSAH)
Keywords: aneurysmal subarachnoid hemorrhage; delayed cerebral ischemia; blood pressure; prognosis
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Target Blood Pressure (Active Comparator): Blood pressure monitoring was initiated immediately upon the patient's return to the intensive care unit (ICU) postoperatively, followed by randomization. Blood pressure management was guided by systolic blood pressure (SBP) measurements, with physicians encouraged to adjust therapy based on institutional protocols and clinical judgment. For SBP <120 mmHg, intravenous crystalloid or colloid fluid resuscitation was prioritized. If the target blood pressure was not achieved, norepinephrine infusion was initiated at a minimum dose of 0.1 µg/kg/min and titrated up to a maximum of 0.5 µg/kg/min to maintain SBP between 120-160 mmHg (<160 mmHg and >120 mmHg). For SBP >160 mmHg, intravenous or oral antihypertensive drugs were administered to reduce and maintain SBP within the 120-160 mmHg range. For SBP within the range of 120-160 mmHg, standard supportive care was provided.
  Interventions: Other: Blood pressure was regulated within the normal target management range
- Elevated Target Blood Pressure (Experimental): Blood pressure monitoring was initiated immediately upon the patient's return to the intensive care unit (ICU) postoperatively, followed by randomization. Blood pressure management was guided by systolic blood pressure (SBP) measurements, with physicians encouraged to adjust therapy based on institutional protocols and clinical judgment. For SBP <160 mmHg, intravenous crystalloid or colloid fluid resuscitation was prioritized. If the target blood pressure was not achieved, norepinephrine infusion was initiated at a minimum dose of 0.1 µg/kg/min and titrated up to a maximum of 0.5 µg/kg/min to maintain SBP between 160-180 mmHg (≤160 mmHg and ≥120 mmHg). For SBP >180 mmHg, intravenous or oral antihypertensive drugs were administered to reduce and maintain SBP within the 160-180 mmHg range. For SBP within the range of 160-180 mmHg, standard supportive care was provided.
  Interventions: Other: Blood pressure was regulated within the elevated target management range

INTERVENTIONS:
Other: Blood pressure was regulated within the normal target management range — Blood pressure monitoring was initiated immediately upon the patient's return to the intensive care unit (ICU) postoperatively, followed by randomization. Blood pressure management was guided by systolic blood pressure (SBP) measurements, with physicians encouraged to adjust therapy based on institutional protocols and clinical judgment. For SBP <120 mmHg, intravenous crystalloid or colloid fluid resuscitation was prioritized. If the target blood pressure was not achieved, norepinephrine infusion was initiated at a minimum dose of 0.1 µg/kg/min and titrated up to a maximum of 0.5 µg/kg/min to maintain SBP between 120-160 mmHg (<160 mmHg and >120 mmHg). For SBP >160 mmHg, intravenous or oral antihypertensive drugs were administered to reduce and maintain SBP within the 120-160 mmHg range. For SBP within the range of 120-160 mmHg, standard supportive care was provided.
  Other Names: normal target blood pressure management
  Arms: Normal Target Blood Pressure
Other: Blood pressure was regulated within the elevated target management range — Blood pressure monitoring was initiated immediately upon the patient's return to the intensive care unit (ICU) postoperatively, followed by randomization. Blood pressure management was guided by systolic blood pressure (SBP) measurements, with physicians encouraged to adjust therapy based on institutional protocols and clinical judgment. For SBP <160 mmHg, intravenous crystalloid or colloid fluid resuscitation was prioritized. If the target blood pressure was not achieved, norepinephrine infusion was initiated at a minimum dose of 0.1 µg/kg/min and titrated up to a maximum of 0.5 µg/kg/min to maintain SBP between 160-180 mmHg ( ≥160 mmHg and ≤120 mmHg). For SBP >180 mmHg, intravenous or oral antihypertensive drugs were administered to reduce and maintain SBP within the 120-160 mmHg range. For SBP within the range of 160-180 mmHg, standard supportive care was provided.
  Other Names: elevated target blood pressure
  Arms: Elevated Target Blood Pressure

SUMMARY:
The goal of this clinical trial is to learn if elevating postoperative blood pressure works to improve prognosis in aneurysmal subarachnoid hemorrhage (aSAH) patients. The main questions it aims to answer are:

Does elevating postoperative blood pressure can improve the prognosis of aSAH ? What safety problems do participants have when received elevating blood pressure measurement?

Participants will:

Receive elevating or lowering blood pressure therapy in 72 hours after randomization, in order to maintain blood pressure within predefined target ranges Receive follow-up at 30 days, 90 days, and 180 days after randomization

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged 18-75 years;

  2) Patients who underwent clipping or endovascular intervention within 72 hours post-ictus;

  3) Intracranial aneurysm diagnosis confirmed by operating surgeons (including neurosurgeons or neurointerventionalists) through imaging findings, intraoperative visualization, or angiography, with subarachnoid hemorrhage (SAH) attributable to the ruptured aneurysm lesion (verified via imaging, xanthochromic cerebrospinal fluid, or intraoperative observation);

  4) Hunt-Hess grade 1-4 at onset;

Exclusion Criteria:

* 1) Presence of untreated intracranial aneurysms with rupture risk;

  2) Moderate-to-severe cerebral vasospasm confirmed by pre-enrollment digital subtraction angiography (DSA), transcranial Doppler (TCD), or computed tomography angiography (CTA);

  3) Intracranial massive hematoma (e.g., volume >30 mL with midline shift >5 mm) causing severe cerebral herniation, as evidenced by admission CT or other imaging modalities;

  4) Prior cranial neurosurgery for other central nervous system disorders;

  5) Comorbid major systemic diseases or multi-organ dysfunction with life expectancy <1 year, potentially compromising study implementation or follow-up observations;

  6) Poorly controlled hypertension despite regular antihypertensive medication (e.g., systolic blood pressure >160 mmHg during pharmacotherapy);

  7) Pre-onset modified Rankin Scale (mRS) score >2 points, indicating disability from other causes;

  8) Intraoperative major complications including but not limited to massive cerebral hemorrhage, hypovolemic shock, or malignant brain swelling;

  9) Anticipated inability to complete scheduled follow-up assessments within 180 days;

  10) Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | Patients received follow-up through telephone consultations or outpatient appointments in the 180 days after randomization. The functional outcome was assessed by the mRS at 90 days post-discharge. mRS 0-2 was considered as favorable clinical outcome.
  The modified Rankin Scale (mRS), a scale ranging from 0 (no symptoms) to 6 (death), is a precise and effective tool to assess the functional outcome of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
To protect patient privacy, the decision was made not to share the data.

REFERENCES:
- [Background] Marbacher S, Neuschmelting V, Andereggen L, Widmer HR, von Gunten M, Takala J, Jakob SM, Fandino J. Early brain injury linearly correlates with reduction in cerebral perfusion pressure during the hyperacute phase of subarachnoid hemorrhage. Intensive Care Med Exp. 2014 Dec;2(1):30. doi: 10.1186/s40635-014-0030-1. Epub 2014 Nov 30. PMID 26266927
- [Background] Tagami T, Kuwamoto K, Watanabe A, Unemoto K, Yokobori S, Matsumoto G, Igarashi Y, Yokota H; SAH PiCCO Study Group. Effect of triple-h prophylaxis on global end-diastolic volume and clinical outcomes in patients with aneurysmal subarachnoid hemorrhage. Neurocrit Care. 2014 Dec;21(3):462-9. doi: 10.1007/s12028-014-9973-z. PMID 24865266
- [Background] Wang J, Lin F, Zeng M, Liu M, Zheng M, Ren Y, Li S, Yang X, Chen Y, Chen X, Sessler DI, Peng Y. Intraoperative blood pressure and cardiac complications after aneurysmal subarachnoid hemorrhage: a retrospective cohort study. Int J Surg. 2024 Feb 1;110(2):965-973. doi: 10.1097/JS9.0000000000000928. PMID 38016131
- [Background] Shah VA, Gonzalez LF, Suarez JI. Therapies for Delayed Cerebral Ischemia in Aneurysmal Subarachnoid Hemorrhage. Neurocrit Care. 2023 Aug;39(1):36-50. doi: 10.1007/s12028-023-01747-9. Epub 2023 May 25. PMID 37231236
- [Background] Minhas JS, Moullaali TJ, Rinkel GJE, Anderson CS. Blood Pressure Management After Intracerebral and Subarachnoid Hemorrhage: The Knowns and Known Unknowns. Stroke. 2022 Apr;53(4):1065-1073. doi: 10.1161/STROKEAHA.121.036139. Epub 2022 Mar 8. PMID 35255708